CLINICAL TRIAL: NCT00819052
Title: An Open Label, Phase IIIb, Randomised Parallel Group Study to Assess the Efficacy and Safety of Switching HIV-1 Infected Patients Successfully Treated With a Nevirapine IR Based Regiment to Nevirapine XR 400 mg QD or Remaining on Nevirapine IR 200 mg BID Based Program
Brief Title: Switching Nevirapine Immediate Release( IR) Based Regimen to Nevirapine Extended Release (XR) Based Regimen in Human Immunodeficiency Virus One (HIV-1) Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1526; 2008-004681-55 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (2):
- NVP IR (Active Comparator): 200 mg orally twice a day (po BID)
  Interventions: Drug: Nevirapine XR; Drug: Nevirapine IR
- NVP XR (Experimental): 400 mg orally once a day (po QD)
  Interventions: Drug: Nevirapine XR

INTERVENTIONS:
Drug: Nevirapine XR — Nevirapine XR
  Arms: NVP IR
Drug: Nevirapine XR — Nevirapine extended release
  Arms: NVP XR
Drug: Nevirapine IR — Nevirapine Immediate Release
  Arms: NVP IR

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of nevirapine extended release (NVP XR) based regimen for HIV-1 infected patients who were receiving nevirapine immediate release (NVP IR) based regimen for at least 18 prior weeks of therapy.

ELIGIBILITY:
Inclusion criteria:

HIV infected subjects treated with a Viramune based regimen.

A subject that meets the following inclusion criteria will be eligible for participation in this study:

1. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation.
2. HIV-1 infected males or females of at least 18 years.
3. Treatment with Viramune regimen for at least the preceding 18 weeks.
4. Background therapy with lamivudine/ abacavir(3TC/ABC) (Kivexa® in EU; Epzicom in US), emtricitabine/tenofovir( FTC/TDF) (Truvada) or lamivudine/zidovudine 3TC/AZT (Combivir®).
5. An HIV viral load < 50 copies/mL in preceding 3 months.
6. An HIV viral load of < 50 copies/mL at screening (Visit 1).
7. Acceptable screening laboratory values that indicate adequate baseline organ function with the following exceptions: alanine aminotrnasferase (ALT) and asparatate aminotransferase (AST) < 2.5 × upper limit of normal (ULN) Division of Acquired Immunodeficiency Syndrome (DAIDS Grade 1).
8. Willingness to abstain from ingesting medications that are listed as contraindicated in the Summary of Product Characteristics (SPC) or package insert (or PI) or Investigator's Brochure during the study.
9. Karnofsky performance score of < 70

Exclusion criteria:

Subjects who meet one or more of the following criteria will be excluded from the study:

1. Current treatment with an HIV protease inhibitor
2. Participation in another trial or use of an investigational medicine within two months prior to Day 1 of this study
3. Female patients of child-bearing potential who:

   1. Have a positive serum pregnancy test at screening.
   2. Are breast feeding.
   3. Are planning to become pregnant
   4. Are not willing to use a double-barrier methods (simultaneous use of two different methods such as diaphragm with spermicidal substance and condom) of contraception, or require ethinyl estradiol administration. Barrier methods of contraception include diaphragm with spermicidal substance, condom for females, cervical caps and condoms..
4. Laboratory parameters > DAIDS grade 2 Coagulation prothrombin time (PT), partial thromboplastin time (PTT), International Normalized ratio (INR) Hematology (absolute platelets, white blood cells (WBC), absolute neutrophil count, hemoglobin) Biochemistry (total bilirubin, amylase, serum creatinine, fasting glucose, lactate, alkaline phosphatase)
5. Laboratory parameters > DAIDS grade 3 Total triglycerides (total cholesterol no restriction)
6. Hypersensitivity to any ingredients of the test products
7. Active drug abuse or chronic alcoholism.
8. Hepatic cirrhosis stage Child-Pugh B or C
9. History of severe or acute illness within 60 days prior to Day 1, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the trial
10. Inability to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (39):
- United States (11):
  - 1100.1526.1012 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1526.1014 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1526.1011 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1100.1526.1013 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1100.1526.1001 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1526.1004 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1526.1006 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1100.1526.1002 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1100.1526.1005 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 1100.1526.1003 Boehringer Ingelheim Investigational Site, Berkley, Michigan
  - 1100.1526.1007 Boehringer Ingelheim Investigational Site, Austin, Texas
- France (9):
  - 1100.1526.3306A Boehringer Ingelheim Investigational Site, Bobigny
  - 1100.1526.3311A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1100.1526.3307A Boehringer Ingelheim Investigational Site, La Roche-sur-Yon
  - 1100.1526.3312A Boehringer Ingelheim Investigational Site, Le Kremlin-Bicêtre
  - 1100.1526.3301A Boehringer Ingelheim Investigational Site, Lyon
  - 1100.1526.3310A Boehringer Ingelheim Investigational Site, Marseille
  - 1100.1526.3308A Boehringer Ingelheim Investigational Site, Montpellier
  - 1100.1526.3302A Boehringer Ingelheim Investigational Site, Nantes
  - 1100.1526.3304A Boehringer Ingelheim Investigational Site, Nice
- Germany (15):
  - 1100.1526.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1526.4903 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1526.4904 Boehringer Ingelheim Investigational Site, Bochum
  - 1100.1526.4905 Boehringer Ingelheim Investigational Site, Bonn
  - 1100.1526.4907 Boehringer Ingelheim Investigational Site, Cologne
  - 1100.1526.4914 Boehringer Ingelheim Investigational Site, Cologne
  - 1100.1526.4906 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1100.1526.4909 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1100.1526.4908 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1526.4901 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1100.1526.4910 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1526.4911 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1526.4912 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1526.4913 Boehringer Ingelheim Investigational Site, Hanover
  - 1100.1526.4915 Boehringer Ingelheim Investigational Site, München
- United Kingdom (4):
  - 1100.1526.4403 Boehringer Ingelheim Investigational Site, London
  - 1100.1526.4405 Boehringer Ingelheim Investigational Site, London
  - 1100.1526.4404 Boehringer Ingelheim Investigational Site, Manchester
  - 1100.1526.4402 Boehringer Ingelheim Investigational Site, Tooting, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients were randomized, but have not been treated. They were excluded from the treated set.
Groups:
- Nevirapine Immediate Release (NVP IR): Nevirapine immediate release 200 mg tablets given twice daily
- Nevirapine Extended Release (NVP XR): Nevirapine extended release 400 mg tablets given once daily
Period: Overall Study
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Started | 148 | 295
Completed | 142 | 281
Not Completed | 6 | 14
Not completed — Adverse Event | 0 | 5
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Pregnancy | 1 | 2
Not completed — Death or events leading to death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR) | Total
Number analyzed (Participants) | 148 | 295 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.8) | 47.3 (9.6) | 47.4 (9.7)
Age, Customized [Number; unit: participants]
  18 to < 41 years | 36 | 70 | 106
  41 to < 56 years | 79 | 168 | 247
  56 to < 65 years | 24 | 38 | 62
  65 years or more | 9 | 19 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 49 | 69
  Male | 128 | 246 | 374
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 5 | 5
  Black | 14 | 20 | 34
  White | 134 | 270 | 404
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic / Latino | 132 | 269 | 401
  Not Hispanic / Latino | 16 | 26 | 42
Region of Enrollment [Number; unit: participants]
  North America | 46 | 98 | 144
  Europe | 102 | 197 | 299
Smoking History [Number; unit: participants]
  Never smoked | 68 | 131 | 199
  Ex-smoker | 37 | 67 | 104
  Current smoker | 43 | 97 | 140
Alcohol Status [Number; unit: participants]
  Non drinker | 44 | 75 | 119
  Drinks - no interfere with trial | 103 | 214 | 317
  Drinks - could interfere with trial | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Virologic Response at Week 24 Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Primary endpoint was the number of patients with a sustained virologic response through week 24
Time Frame: week 24
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 137 | 276
  Non responder | 11 | 19
Statistical Analysis 1: Comparison: Nevirapine Immediate Release (NVP IR) vs Nevirapine Extended Release (NVP XR); Test type: Non-Inferiority or Equivalence — Non-inferiority of nevirapine XR to nevirapine IR was established if the lower bound of the confidence interval was greater than -12%; Cochran's statistic; Cochran's statistic = 1.0, 95% CI [-4.3 to 6.2] — Weighted treatment difference and corresponding variance were calculated based on Cochran's statistic

2. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 400 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 2
Time Frame: week 2
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 148 | 292
  Non responder | 0 | 3

3. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 400 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 4
Time Frame: week 4
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 146 | 291
  Non responder | 2 | 4

4. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 400 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 8
Time Frame: week 8
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 146 | 290
  Non responder | 2 | 5

5. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 400 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 12
Time Frame: week 12
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 143 | 289
  Non responder | 5 | 6

6. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 400 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 24
Time Frame: week 24
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Responder | 140 | 285
  Non responder | 8 | 10

7. Secondary Outcome: Kaplan-Meier Estimates of the Proportions of Patients Without Loss of Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Time Frame: week 0 to 24
Population: as for baseline characteristics
Measure: Number; unit: proportion of participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
proportion of participants
  Interval Week 0 to <2 | 1 | 1
  Interval Week 2 to <4 | 1 | 0.986
  Interval Week 4 to <8 | 0.993 | 0.98
  Interval Week 8 to <12 | 0.973 | 0.973
  Interval Week 12 to <16 | 0.959 | 0.966
  Interval Week 16 to <20 | 0.946 | 0.953
  Interval Week 20 to <24 | 0.946 | 0.946
  Interval Week 24 to <28 | 0.946 | 0.942

8. Secondary Outcome: Summary of CD4 Count (Cells/Cubic Millimeter) at Baseline, Full Analysis Set Population
Time Frame: week 0
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 147 | 295
cells/cubic millimeter | 569.7 (215.6) | 557.7 (213.2)

9. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 2, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 2
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline and week 2.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 141 | 280
cells/cubic millimeter | 3.7 (115.2) | -4.7 (107.7)

10. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 4, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 4
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline and week 4.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 137 | 271
cells/cubic millimeter | 0.8 (110.8) | -15.4 (114.1)

11. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 8, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 8
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline and week 8.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 139 | 281
cells/cubic millimeter | -18.6 (122.9) | -24.4 (117.6)

12. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 12, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 12
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline and week 12.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 139 | 283
cells/cubic millimeter | 22.3 (152.9) | -10.2 (118.5)

13. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 24, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 24
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants who had CD4 count at baseline and week 24.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 142 | 282
cells/cubic millimeter | 50.4 (162.8) | 45.7 (137.6)

14. Secondary Outcome: Comparison of CD4 Count (Cells/Cubic Millimeter) Change From Baseline at Week 24, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 24
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment.The population was restricted to participants who had CD4 count at baseline and week 24.
Measure: Least Squares Mean (Standard Error); unit: cells/cubic millimeter
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 142 | 282
cells/cubic millimeter | 50.74 (12.7072) | 46.10 (9.2053)
Statistical Analysis 1: Comparison: Nevirapine Immediate Release (NVP IR) vs Nevirapine Extended Release (NVP XR); Test type: Superiority or Other; p = 0.7587, ANCOVA; Means adjusted for background ARV (Antiretroviral) stratum; Mean Difference (Final Values) = -4.64, 95% CI [-34.34 to 25.05]

15. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 48
Time Frame: week 48
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants present at week 48.
Measure: Number; unit: participants
Groups:
- Nevirapine (NVP) IR / NVP XR: Nevirapine IR during first 48 weeks then switched to NVP XR
- Nevirapine IR After Week 48: Patient remained on NVP IR after week 48
- Nevirapine XR After Week 48: Patient remained on NVP XR after week 48
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 130 | 12 | 276
participants
  Responder | 125 | 11 | 268
  Non responder | 5 | 1 | 8

16. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 60
Time Frame: week 60
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 60.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 130 | 12 | 274
participants
  Responder | 122 | 9 | 253
  Non responder | 8 | 3 | 21

17. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 72
Time Frame: week 72
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 72.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 130 | 9 | 271
participants
  Responder | 124 | 9 | 265
  Non responder | 6 | 0 | 6

18. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 84
Time Frame: week 84
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 84.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 125 | 8 | 268
participants
  Responder | 118 | 7 | 244
  Non responder | 7 | 1 | 24

19. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 96
Time Frame: week 96
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 96.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 124 | 9 | 263
participants
  Responder | 117 | 9 | 242
  Non responder | 7 | 0 | 21

20. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 108
Time Frame: week 108
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 108.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 125 | 9 | 260
participants
  Responder | 119 | 8 | 247
  Non responder | 6 | 1 | 13

21. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 120
Time Frame: week 120
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 120.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 121 | 8 | 258
participants
  Responder | 112 | 7 | 235
  Non responder | 9 | 1 | 23

22. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 132
Time Frame: week 132
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 132.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 121 | 7 | 252
participants
  Responder | 115 | 6 | 238
  Non responder | 6 | 1 | 14

23. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response through week 144
Time Frame: week 144
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at week 144.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 121 | 7 | 250
participants
  Responder | 115 | 7 | 238
  Non responder | 6 | 0 | 12

24. Secondary Outcome: Number of Participants With Virologic Response Using Lower Limit of Quantification (LLOQ) = 50 Copies/mL, Full Analysis Set Population
Description: Endpoint was the number of patients with a sustained virologic response at their last available visit
Time Frame: last available visit, up to 144 weeks
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to patients present at last visit (up to 144 weeks).
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 130 | 13 | 276
participants
  Responder | 121 | 11 | 261
  Non responder | 9 | 2 | 15

25. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 48, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 48
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 48.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 126 | 11 | 267
cells/cubic millimeter | 77.8 (142.8) | 139.8 (126.9) | 52.7 (143.5)

26. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 60, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 60
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 60.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 126 | 12 | 273
cells/cubic millimeter | 51.1 (138.1) | 11.5 (138.4) | 55.1 (136.5)

27. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 72, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 72
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 72.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 126 | 9 | 265
cells/cubic millimeter | 61.3 (128.6) | 77.9 (109.5) | 67.4 (141.5)

28. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 84, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 84
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 84.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 123 | 8 | 265
cells/cubic millimeter | 80.3 (156.5) | 134.6 (214.2) | 55.0 (130.9)

29. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 96, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 96
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 96.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 120 | 8 | 239
cells/cubic millimeter | 55.1 (156.7) | 55.4 (80.7) | 60.2 (130.3)

30. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 108, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 108
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 108.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 124 | 8 | 256
cells/cubic millimeter | 72.4 (160.4) | 117.4 (151.3) | 73.5 (151.0)

31. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 120, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 120
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 120.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 119 | 8 | 258
cells/cubic millimeter | 79.5 (168.4) | 90.0 (151.0) | 66.6 (182.3)

32. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 132, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 132
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 132.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 120 | 7 | 252
cells/cubic millimeter | 58.8 (153.6) | 124.8 (158.7) | 70.8 (146.7)

33. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Week 144, Observed Cases, Full Analysis Set Population
Time Frame: baseline, week 144
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and week 144.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 120 | 7 | 250
cells/cubic millimeter | 85.3 (151.6) | 205.6 (388.6) | 82.7 (157.4)

34. Secondary Outcome: Change From Baseline in CD4 Count (Cells/Cubic Millimeter) at Last Available Visit, Observed Cases, Full Analysis Set Population
Time Frame: baseline, last available visit (up to 144 weeks)
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants with CD4 counts at baseline and last visit (up to 144 weeks).
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 129 | 13 | 276
cells/cubic millimeter | 71.9 (157.1) | 165.9 (302.5) | 80.9 (163.5)

35. Secondary Outcome: Proportion of Virologic Response (Viral Load <400 Copies/mL) Trough Week 144
Description: Endpoint was the number of patients with a sustained virologic response through week 144
Time Frame: week 144
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment. The population was restricted to participants present at week 144.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 121 | 7 | 250
participants
  Responder | 121 | 7 | 250
  No Responder | 0 | 0 | 0

36. Secondary Outcome: Change From Baseline in VL (HIV-1 Viral Load) at Each Visit
Time Frame: week 48, 60, 72, 84, 96, 108, 120, 132, 144, last available visit
Population: Full Analysis Set (FAS) includes all participants randomized to treatment and confirmed to have taken at least one dose of treatment, Observed Cases.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Nevirapine (NVP) IR / NVP XR | Nevirapine IR After Week 48 | Nevirapine XR After Week 48
Number analyzed (Participants) | 130 | 13 | 276
copies/mL
  week 48 (N=130, 12, 275) | 48.4 (536.9) | 58.4 (202.3) | -4.3 (67.6)
  week 60 (N=130, 12, 274) | 11004.4 (125415) | 94.1 (218.5) | -1.8 (69.4)
  week 72 (N=129, 9, 271) | 1747.0 (19806) | 0.0 (0.0) | -4.9 (68.2)
  week 84 (N=125, 8, 268) | 2798.8 (31301) | 4.1 (11.7) | 4140.1 (67801)
  week 96 (N=124, 9, 263) | 0.2 (17.7) | 0.0 (0.0) | 168.4 (1974.7)
  week 108 (N=125, 8, 260) | 53.1 (574.2) | 0.0 (0.0) | -3.5 (70.6)
  week 120 (N=121, 8, 257) | 3.5 (42.7) | 0.4 (1.1) | -2.3 (71.0)
  week 132 (121, 7, 252) | 10.2 (78.7) | 4.0 (10.6) | -1.8 (79.0)
  week 144 (N=121, 7, 250) | 1.0 (24.5) | 0.0 (0.0) | -4.6 (70.9)
  last available visit(N=130,13,276) | 4472.6 (36357) | 86.4 (211.0) | 4103.2 (66822)

37. Secondary Outcome: Changes in Safety Parameters Related to Treatment
Description: Occurence of investigations related to treatment
Time Frame: until week 144
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  Alanine aminotransferase increased | 1 | 4
  Aspartate aminotransferase increased | 0 | 2
  Blood amylase increased | 1 | 0
  Blood triglycerides increased | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 2
  Lipase increased | 1 | 0
  Liver function test abnormal | 1 | 0
  Blood glucose increased | 0 | 1
  Blood lacate dehydrogenase increased | 0 | 1
  Neutrophil count decreased | 0 | 1
  Transaminases increased | 0 | 1

38. Secondary Outcome: Occurence of Rashes
Description: drug-related rashes by severity
Time Frame: 144 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  rash Grade 1 mild | 0 | 1
  rash Grade 2 moderate | 0 | 1
  rash Grade 3 severe | 0 | 0
  rash Grade 4 potential life-threatening | 0 | 0

39. Secondary Outcome: Occurence of Hepatic Events
Time Frame: 144 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants | 0 | 1

40. Secondary Outcome: New AIDS or AIDS-related Progression Event or Death
Time Frame: 144 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
participants
  new AIDS or AIDS related progression | 1 | 2
  death | 2 | 2

41. Secondary Outcome: Time to Loss of Virologic Response
Description: Kaplan-Meier Estimates of time to loss of virologic response defined as the time between the start of treatment and the time of treatment failure, up to and including the time when the last patient was on treatment for 48 weeks.
Time Frame: 48 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
days | 393 [393 to 406] | 391 [377 to 423]

42. Secondary Outcome: Genotypic Resistance Associated With Virologic Failure
Description: Genotypic resistance associated with virologic failure.
  This endpoint was not analysed due to lack of data.
Time Frame: 48 weeks
Population: All patients in the treated set who experienced virologic failure.
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Trough Plasma Concentration
Description: Trough plasma concentrations of Nevirapine at steady state after multiple oral administrations of Nevirapine treatments from day 1 (visit 2) to week 48 (visit 9).
Time Frame: Day 1 to week 48
Population: All patients with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Number analyzed (Participants) | 148 | 295
ng/mL
  Day 1 (N=146, 0) | 3720 (65.4) | NA (NA) — No data was available at this time point
  Week 2 (N=107, 229) | 3650 (38.1) | 3270 (57.6)
  Week 4 (N=103, 234) | 3720 (36.6) | 3230 (49.0)
  Week 8 (N=110, 225) | 4080 (38.2) | 3650 (46.1)
  Week 12 (N=103, 223) | 4170 (41.1) | 3590 (50.2)
  Week 24 (N=103, 212) | 4080 (36.9) | 3750 (41.8)
  Week 36 (N=103, 215) | 4370 (40.6) | 3930 (41.5)
  Week 48 (N=101, 213) | 3960 (41.8) | 3650 (45.0)

ADVERSE EVENTS:
Time Frame: 144 weeks
Arm/Group | Nevirapine Immediate Release (NVP IR) | Nevirapine Extended Release (NVP XR)
Serious Adverse Events (participants affected / at risk) | 33/148 | 73/295
Other Adverse Events (participants affected / at risk) | 110/148 | 244/295
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine Immediate Release (NVP IR) (N=148) | Nevirapine Extended Release (NVP XR) (N=295)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Pericarditis (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 2
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Dysplasia (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2
Chronic sinusitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 1
Shigella infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood lactic acid increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem ischaemia (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine Immediate Release (NVP IR) (N=148) | Nevirapine Extended Release (NVP XR) (N=295)
Conjunctivitis (Eye disorders) | 8 | 11
Diarrhoea (Gastrointestinal disorders) | 20 | 62
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 16
Nausea (Gastrointestinal disorders) | 4 | 20
Fatigue (General disorders) | 9 | 30
Bronchitis (Infections and infestations) | 24 | 49
Gastroenteritis (Infections and infestations) | 12 | 16
Herpes zoster (Infections and infestations) | 3 | 15
Nasopharyngitis (Infections and infestations) | 25 | 74
Pharyngitis (Infections and infestations) | 10 | 16
Sinusitis (Infections and infestations) | 20 | 33
Syphilis (Infections and infestations) | 7 | 24
Upper respiratory tract infection (Infections and infestations) | 21 | 35
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 40
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 16
Headache (Nervous system disorders) | 13 | 31
Depression (Psychiatric disorders) | 10 | 33
Insomnia (Psychiatric disorders) | 9 | 22
Sleep disorder (Psychiatric disorders) | 4 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 36
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 16
Eczema (Skin and subcutaneous tissue disorders) | 1 | 18
Hypertension (Vascular disorders) | 15 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.